CLINICAL TRIAL: NCT06486610
Title: Inhalation With Toy Figure and Sound Insulated Nebulizer Effect of Treatment on Children's Fear and Anxiety Levels and Physiological Parameters: Randomized Controlled Study
Brief Title: Effect of Inhalation Therapy on Children's Fear and Anxiety Levels and Physiological Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Mehtap METİN KARAASLAN, Study Director, Recep Tayyip Erdogan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1528/TSA-2023-1528
Record Dates: First submitted 2024-05-03; First posted 2024-07-03 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Anxiety and Fear
Keywords: child; nebulizer; fear; anxiety; therapeutic play
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group: Routine clinical practice (No Intervention): Fear, Emotional Indicators and Physiological Parameters in Children
- Therapeutic play: Fish-shaped nebulizer and fish-shaped toy (Experimental): Fear, Emotional Indicators and Physiological Parameters in Children
  Interventions: Behavioral: Fish-shaped nebulizer and fish-shaped toy
- silent nebulizer (Experimental): Fear, Emotional Indicators and Physiological Parameters in Children
  Interventions: Device: Silent nebulizer

INTERVENTIONS:
Behavioral: Fish-shaped nebulizer and fish-shaped toy — In order to reduce the child's fear and anxiety, it is planned to apply inhalation therapy using a nebulizer with a red fish figure and an amigurumi toy with a red fish figure.
  Arms: Therapeutic play: Fish-shaped nebulizer and fish-shaped toy
Device: Silent nebulizer — It is planned to apply inhalation therapy using a silent nebulizer to reduce the child's fear and anxiety.
  Arms: silent nebulizer

SUMMARY:
The research was planned as a randomized controlled study. Between July 2023 and July 2025, he was hospitalized in the pediatric emergency department of Recep Tayyip Erdogan University Training and Research Hospital and was treated with a nebulizer. It includes children aged 3-6 and their mothers receiving treatment. The sample of the research will consist of 120 children and their mothers who applied to the pediatric emergency department between the specified dates and met the inclusion criteria and volunteered to participate in the research. "Introductory Information Form", "Child Fear Scale", "Emotional Indicators Scale in Children", "Physiological Parameter Tracking Form" will be used to collect data. "Nebulizer with Toy Figure", "Sound Insulated (Silent) Nebulizer" and "Toy with Fish Figure" will be used as research materials.

DETAILED DESCRIPTION:
The research was planned as a randomized controlled study. Between July 2023 and July 2025, he was hospitalized in the pediatric emergency department of Recep Tayyip Erdogan University Training and Research Hospital and was treated with a nebulizer. It includes children aged 3-6 and their mothers receiving treatment. The sample of the research will consist of 120 children and their mothers who applied to the pediatric emergency department between the specified dates and met the inclusion criteria and volunteered to participate in the research. "Introductory Information Form", "Child Fear Scale", "Emotional Indicators Scale in Children", "Physiological Parameter Tracking Form" will be used to collect data. "Nebulizer with Toy Figure", "Sound Insulated (Silent) Nebulizer" and " Toy with Fish Figure" will be used as research materials.

Data Collection:

Data for the study will be obtained through face-to-face interviews. Initially, children in the groups using either a toy-figured nebulizer or a Sound-Insulated (Silent) Nebulizer will complete an Introductory Information Form. The physiological parameters of the children will be measured by an experienced nurse in pediatric emergency care 15 minutes before, during the 10th minute of, and 15 minutes after the nebulizer medication application, and recorded on a 'Physiological Parameters Form.' Additionally, the Child Fear Scale and the Emotional Indicators in Children Scale will be administered 15 minutes before, during the 10th minute of, and 15 minutes after the medication application with the toy-figured nebulizer. For the control group, routine inhalation therapy of the service will be applied without any additional intervention. Children in this group will also fill out the Introductory Information Form. Their life signs will be measured similarly by the experienced nurse and recorded on a 'Physical Parameters Form.' The Child Fear Scale and Emotional Indicators in Children Scale will be administered during the 10th minute and 15 minutes after the routine medication application. Due to the nature of the study, blinding during the execution will not be possible; however, to prevent potential bias, measurements will be taken by both the experienced nurse (for physiological parameters, Child Fear Scale, Emotional Indicators in Children Scale) and parents (for Child Fear Scale, Emotional Indicators in Children Scale). Statistical analysis and reporting will be conducted without knowledge of which group is the experimental or control group (coding will be applied).

Data Evaluation:

Data processing and statistical analyses will be performed using Statistical Package for the Social Sciences for Windows 20.0. For measurements not conforming to a normal distribution, non-parametric methods will be utilized. The Kruskal-Wallis H test (χ2-table value) will be used for comparing three or more independent groups. Pearson-χ2 cross-tabulations will be employed to examine the relationships between two qualitative variables. The Spearman correlation coefficient will be used to analyze the relationships between two quantitative variables that do not follow a normal distribution.

Ethical Principles of the Research:

For the execution of the study, official permission has been obtained from the Ethical Committee of the Recep Tayyip Erdogan University Faculty of Medicine. Children eligible for the research group, along with their parents, will be informed about the purpose of the study, and their questions will be answered before obtaining their verbal and written consent. Parents and children will be assured that the data collected during the research will be processed anonymously and confidentially, will not be used outside of this study, and they may withdraw from the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Having a child between the ages of 3-6
* Nebulizer and inhaler treatment will be applied
* The child does not have a mental or neurological disability
* Applying due to respiratory system disease
* The presence of the child's mother during the application period
* Mother and child can speak Turkish
* The mother does not have any obstacle to communication
* Mother's literacy
* Parent and child volunteering to participate in the research.

Exclusion Criteria:

* The child and parent have previously experienced inhalation therapy with a nebulizer.
* The child is hyperthermic (body temperature is 38 C and above)
* The child has pain,
* The child is in the terminal period,
* The parent has a condition that prevents him/her from evaluating the scale (mental disability, etc.).

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Child Fear Scale | one year
  This scale was developed to measure the anxiety levels in children. The facial muscle changes in expressions of fear have been illustrated by a graphic artist based on photographs of frightened faces. The scale can be used by families, children, or researchers to assess children. It presents a scale containing five facial expressions, scored between 0 and 4. A score of 0 indicates no fear or anxiety, while a score of 4 indicates the highest level of fear or anxiety. These are recognized as: "0" neutral expression (no anxiety), "1" very slight fear (very low anxiety), "2" mild fear (mild anxiety), "3" more fear (increased anxiety), "4" the most extreme fear (severe anxiety). This scale can be applied to measure fear and anxiety before and during medical procedures.
Emotional Indicators Scale for Children | one year
  This scale is an easily administered and evaluated tool used to objectively identify emotional responses of children to medical procedures. The emotional indicators on the scale are assessed based on five parameters: facial expression, voice, activity, interaction, and cooperation level. These five parameters are scored from 1 to 5, with the lowest possible score being 5 and the highest being 25. The scale has a Cronbach's alpha reliability coefficient of 0.88. In this study, the scale will be utilized to assess the emotional indicators of children during inhalation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mehtap METİN KARAASLAN, Study Director — Recep Tayyip Erdogan Universİty
Locations (1):
- Recep Tayyip Erdoğan University Faculty of Health Sciences, Rize, Güneysu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No